CLINICAL TRIAL: NCT01485575
Title: Mechanical Properties of the Internal Limiting Membrane and Intraoperative Utility of Brilliant Blue g (Bbg) and Indocyanine Green (Icg) Assisted Chromovitrectomy
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: University of the Italian Switzerland (Other); Clinical Trial Unit, University Hospital Basel, Switzerland (Other); General Hospital Linz (Other); Oftacentro SA (Other)
Responsible Party: Sponsor
Other Study IDs: ILM-AMF2
Record Dates: First submitted 2011-11-28; First posted 2011-12-05 (Estimated); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Macular Edema
Keywords: Chromovitrectomy; Indocyanine green; ICG; Brilliant Blue G; BBG; Trypan blue; TB; Internal limiting membrane; ILM
MeSH Terms: conditions — Macular Edema | interventions — Vitrectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Internal limiting membrane as removed during routine surgery.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Filter use during vitrectomy
  Interventions: Procedure: Use of intraoperative filters in vitrectomy

INTERVENTIONS:
Procedure: Use of intraoperative filters in vitrectomy — During vitrectomy with xenon endoillumination, an orange, green and a yellow filter are applied sequentially to determine which one produces the best contrast behavior of vital dyes
  Other Names: Stellaris PC surgical (Bausch&Lomb surgical,Aliso Viejo,CA)

SUMMARY:
Intravitreal dyes are intended to make the surgical extraction of the Internal limiting membrane (ILM) safer and more complete. However, the search for an adequate vitaly dye is ongoing. The most commonly used vital dye is Indocyanine green (ICG), although it is not approved for intravitreal use and has been associated with ocular toxicity. The reason for its continued popularity seems to be that it stains the ILM better than the approved and less toxic alternative substances Brilliant Blue G (BBG) and Trypan blue (TB). According to anecdotal reports from surgeons, another reason for ICGs popularity may be the fact that it seems to make ILM removal easier. Ultimately, the intention of the investigators research is to identify possible modifications to existing dyes to reach improved intraoperative dye utility combined with a favorable safety profile.

Protocol was amended and approved concerning additional use of basal membrane of deceased donors.

DETAILED DESCRIPTION:
The human retina is a light-sensitive tissue lining the inner surface of the posterior segment of the eye. It is a complex, layered structure containing the photoreceptors and several layers of neurons. Proper retinal function requires a smooth interface between the retina and the adjoining vitreous body (vitreous), a gelatinous and transparent substance occupying the cavity of the posterior ocular segment. The innermost of the retinal layers, a basement membrane called Inner limiting membrane (ILM), represents the boundary between the retina and the vitreous. Excessive contact between the ILM and the vitreous leads to vitreoretinal traction and represents a common cause of ocular pathology: The vitreous adheres to the ILM and shearing forces are conveyed to the retina. Vitreoretinal traction concentrates around the Macula lutea, the small area in the center of the retina which is responsible for central vision. It may be associated with significant visual disturbance as it creates retinal folds, provokes retinal edema and epiretinal metaplastic membranes through the liberation of inflammatory messenger substances and may ultimately result in the formation of macular holes. Macular holes tend to lead to sudden and often complete loss of central vision.

Removal of the vitreous (vitrectomy) may improve vitreoretinal traction, but a complete relief of traction is only achieved if the ILM is removed from the retina in the area around the macula: At the end of vitrectomy, the surgeon grasps the ILM with a fine forceps and carefully peels it off the underlying retinal layers. This procedure is extremely delicate, as the ILM is transparent, extremely thin and in direct contact with highly vulnerable retinal structures. Vital dyes have been employed to make the ILM more visible and because some dyes have been described to improve "grip" of the ILM during its extraction. The most commonly used dye, Indocyanine green (ICG) is not approved for intravitreal use and a discussion on possible toxic side effects is ongoing. The approved alternative substance Brilliant blue G is employed only by a minority of vitreoretinal surgeons. It is our hypothesis, that the popularity of ICG is due to superior staining capacity and a stiffening effect which may make ILM removal easier for the surgeon.

The first goal of this interdisciplinary and translational project, integrating Medical physics, Biomedical engineering, Nanosciences, Biochemistry, Neurobiology, Medical Image analysis and Clinical ophthalmology is to assess the biophysical properties of the ILM and the possible effects of existing dyes in terms of staining behavior and their influence on ILM "grip". In a second step, the project will analyze how new application protocols and the introduction of novel components to the molecular structure of vital dyes can improve staining as well as "ILM-grip" while guaranteeing favorable toxicity profiles Hypotheses

1. A novel "Heavy BBG" (BBG D2O) stains the ILM better than conventional BBG. A replacement of part of the water molecules with Deuterium Oxide (D20) in the BBG solvent increases the dye's specific gravity. After injection into the vitreous, this new preparation (BBG D2O) would collect on the retinal surface, increasing local concentration and retinal exposure. We hypothesize that this alteration of the BBG molecular structure could improve staining properties without compromising its favorable toxicity profile. This new BBG has already been introduced by the manufacturer, but its intraoperative usefulness has not been objectively examined.
2. The use of intraoperative light filters improves the recognizability of the contrasts generated by vital dyes. Most endoillumination lighting systems are equipped with light filters, originally intended to reduce intraoperative light toxicity. Anecdotal reports by numerous surgeons indicate, however, that the use of some filters improves the recognizability of the stained ILM. The green filter is regarded as particularly useful for this purpose. A systematic analysis of the effects of light filters on the usefulness of intravitreal dyes has not been undertaken to date.
3. ICG and TB's photochemical properties improve "ILM grip" through an ILM cross-linking effect resulting in an alteration of ILM material properties. We expect increased intra-operative ILM compressive and tensile stiffness and reduced ILM thickness in Atomic force microscopy examinations, explaining why many surgeons describe facilitated intraoperative manipulation and extraction of the ILM. BBG is not known to dispose of photochemical properties and should not influence ILM material properties.
4. Novel Modified ICG preparation stains equally well but is less toxic An alteration of the molecular structure in a way such that photochemical properties of the substance would be largely eliminated would strongly reduce oxidative stress and retinal toxicity. Synthetization of such a preparation is being prepared by our group. Staining properties are different from the original preparation in that the absorption maximum is shifted towards shorter wavelengths and the staining effect is bluish rather than green. The substance's affinity to the ILM its staining strength and its toxicity have not been studied, to date.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 Years of age
* No other chromovitrectomy in previous 6 months
* Only one of three vitaly dyes used intraoperatively (BBG, ICG or TB)

Exclusion Criteria:

* Previous chromovitrectomy during last 6 months
* Pregnant patients
* Patients under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients treated with Chromovitrectomy at 3 tertiary care hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2011-11; Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
ILM thickness, stiffness and roughness | No further patient contact is required after surgery. Analysis of the specimens may take up to one year
  Measurements under the Atomic force microscope will show wether the use of ICG or BBG influences material properties of the ILM (for example, an increased stiffness may explain a better "grip").

SECONDARY OUTCOMES:
Contrast between the stained ILM and the underlying tissue | No further patient contact is required after surgery. Analysis of the video frames may take up to one year
  Intraoperative videos will be analysed to understand under which circumstances vital dyes produce the best contrast visible to the human eye

CONTACTS AND LOCATIONS:
Overall Officials: Paul B Henrich, MD, Principal Investigator — Oftacentro, Lugano-Paradiso, Switzerland
Locations (3):
- General Hospital Linz, Linz, Austria
- Switzerland (2):
  - St. Gallen Hospital, Sankt Gallen, Canton of St. Gallen
  - Oftacentro, Paradiso, Canton Ticino

IPD SHARING:
Plan to Share IPD: Undecided